CLINICAL TRIAL: NCT06605092
Title: Characterization of Emotional Response Profiles Triggered by a Digital Artwork of Musicalized Impressionist Paintings
Acronym: NeuroArt
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre integre universitaire de sante et de services sociaux du Centre-Sud-de-l'Île-de-Montréal (Other Government)
Responsible Party: Principal Investigator, Olivier Beauchet, MD, PhD, Centre integre universitaire de sante et de services sociaux du Centre-Sud-de-l'Île-de-Montréal
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2025-2242
Record Dates: First submitted 2024-09-13; First posted 2024-09-20 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Anxiety
Keywords: ecoanxiety; art; emotions
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: 2 groups (young adults and older adults), with a 50/50 male/female ratio in each group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Young Adults (Experimental): Adults from 18 to 35 years old
  Interventions: Other: Emotional stimulation
- Elderly (Experimental): Adults aged 65 years ol or more
  Interventions: Other: Emotional stimulation

INTERVENTIONS:
Other: Emotional stimulation — Presentation of the paintings by distinguishing 3 conditions: (1) contemplating each painting (visual stimulation), (2) listening to the original music composed from each painting (auditory stimulation), (3) contemplating and listening to the association of each painting with each specific music (bimodal stimulation)

SUMMARY:
Global warming, progressing at a rapid pace in Canada, is causing severe consequences for ecosystems and human health. Rising temperatures accelerate glacier melting, increase heat waves, and disrupt biodiversity. These environmental changes impact mental health, notably through ecoanxiety, a form of anxiety linked to climate change. Although ecoanxiety is a natural reaction to environmental degradation, it can lead to chronic stress, generalized anxiety, and even depression. Recent studies show that ecoanxiety is increasingly common, especially among young people. In Quebec, 73% of young adults (18-35 years) report experiencing ecoanxiety, with 42% experiencing significant levels. Vulnerable populations, such as Indigenous communities like the Inuit of Nunavik, are particularly affected.

To address ecoanxiety, interventions focused on emotional management and reconnecting with nature are essential. Studies show that outdoor activities such as walking or gardening reduce negative emotions and improve well-being by fostering a connection with nature, thereby increasing resilience to climate change.

Art, especially pictorial art, is emerging as a promising tool in combating ecoanxiety. The World Health Organization (WHO) recognizes the mental health benefits of art, which is not only beneficial for those suffering from mental illness but also for the general population. The Quebec Interministerial Mental Health Action Plan (PAISM) 2022-2026 highlights the promotion of art as a priority in mental health prevention. Among art forms, the contemplation of Impressionist paintings has shown positive effects, generating emotions of serenity and deeper reflection on our relationship with nature. Music therapy also plays a vital role in anxiety management, promoting relaxation and emotional expression.

Music, in particular, has shown promise in reducing ecoanxiety. Listening to music can alleviate anxiety and depression by stimulating the limbic system, which regulates emotions. Music can also modulate physiological stress responses and strengthen personal resilience, enhancing emotional regulation in environmental crises. An innovative approach involves creating music from electrophysiological signals captured from plants, a process known as sonification. This nature-inspired music fosters a deeper connection with the environment, potentially reducing ecoanxiety and increasing resilience.

Emotions, both positive and negative, are central to mental health. According to James Russell's circumplex theory of emotions, they are classified into two dimensions: valence (pleasant or unpleasant) and arousal (energy level). Positive emotions like joy and relaxation promote well-being, while negative emotions, such as anxiety and sadness, have detrimental effects on mental health. Emotional responses manifest through physiological changes, such as increased heart rate and skin conductance. Modern technologies, like functional MRI, allow researchers to observe the brain's activity in areas like the amygdala, responsible for emotional regulation.

Digital technologies have revolutionized the use of art in promoting mental health. Immersive digital interventions, such as apps that allow users to experience art online, have shown positive results. One such app currently in development combines the works of Impressionist painters Claude Monet and Helen McNicoll with music created from plant electrophysiological signals. This digital combination of art and nature offers emotional benefits, promoting well-being in the face of climate challenges.

It is well-established that positive emotions play a crucial role in improving mental health and protecting against ecoanxiety. Research shows that Impressionist paintings and music can generate positive emotions. This study hypothesizes that (1) observing and listening to musicalized paintings can generate positive emotions, (2) the emotional effect is stronger when both stimuli are combined, and (3) these emotions vary with age.

DETAILED DESCRIPTION:
Global warming, which is progressing at a particularly rapid pace in Canada, is having a multitude of serious consequences for ecosystems and human health. Rising temperatures are accelerating the melting of glaciers, increasing the frequency of heat waves and profoundly disrupting biodiversity. These environmental upheavals also have repercussions on mental health, notably through ecoanxiety, a form of anxiety linked to climate change. Although ecoanxiety is a natural reaction to environmental degradation, it can lead to chronic stress, generalized anxiety and, in some cases, depression. Recent studies have shown that this form of anxiety is increasingly common, particularly among younger generations. In Quebec, for example, 73% of young adults aged 18 to 35 declare themselves to be ecoanxious, with 42% claiming to experience significant ecoanxiety. The psychological effects are even more pronounced among vulnerable populations, such as young people, aboriginal peoples, or those living in regions severely affected by climate change, like the Inuit of Nunavik.

To combat this form of anxiety, it is essential to implement interventions focused on managing emotions and reconnecting with nature. Studies show that outdoor activities such as walking or gardening can reduce negative emotions and improve well-being. These practices help individuals to reconnect with the environment, strengthening their resilience in the face of climate change.

At the same time, art, particularly pictorial art, is emerging as a promising solution to eco-anxiety. The World Health Organization (WHO) recognizes the benefits of art for mental health, pointing out that artistic activities are not only beneficial for sufferers, but also for people in general, whatever their age. The Plan québécois d'action interministériel en santé mentale (PAISM) 2022-2026 includes the promotion of art as a priority in the prevention and promotion of mental health. Among art forms, the contemplation of pictorial works, particularly those by Impressionist painters, has been shown to be effective in generating positive emotions. These paintings, often centered on nature, create a sense of serenity and beauty, encouraging deeper reflection on our relationship with the natural world. In addition to pictorial art, music is also recognized for its positive impact on anxiety management. Music therapy, for example, helps to reduce stress and anxiety, by promoting relaxation and emotional expression.

Music, in particular, plays an important role in combating ecoanxiety. Research shows that listening to music can alleviate symptoms of anxiety and depression by stimulating the limbic system, the area of the brain responsible for emotions. In addition, music can modulate physiological responses to stress and strengthen personal resilience, contributing to better emotional regulation in the face of environmental crises. An innovative approach in this field involves creating music from electrophysiological signals captured on plants. This technique, known as sonification, transforms these signals into sounds, offering music inspired by nature. By fostering a deeper connection with the environment, this type of music could reduce eco-anxiety and increase resilience in the face of ecological challenges.

Emotions, both positive and negative, play a central role in mental health. According to James Russell's circumplex theory of emotions, emotions can be classified into two dimensions: valence (pleasant or unpleasant) and arousal (energy level). Positive emotions with high arousal, such as joy, or low arousal, such as relaxation, are beneficial to well-being. On the other hand, negative emotions, whether high arousal (such as anxiety) or low arousal (such as sadness), can have deleterious effects on mental health. These emotional responses manifest themselves through neurophysiological changes, such as increased heart rate or changes in skin conductance. Modern technologies, such as functional magnetic resonance imaging (fMRI), make it possible to explore these responses by observing the activity of brain areas involved in emotion management, such as the amygdala or the prefrontal cortex.

Finally, digital technology has revolutionized the way art can be used to promote mental health. Immersive digital interventions, such as apps that allow people to contemplate works of art online, have shown promising results. An application currently under development, for example, offers immersion in the work of Impressionist painters such as Claude Monet or Helen McNicoll, combined with music created from the sonification of electrophysiological signals from plants. This combination of art and nature, via digital technology, maximizes emotional benefits and promotes sustainable well-being in the face of climate challenges.

RESEARCH HYPOTHESIS It is now proven that positive emotions play a crucial role in promoting and improving mental health, contributing to enhanced well-being. Some research suggests that positive emotions may also play a protective role against the negative consequences of ecoanxiety. So, while ecoanxiety is mainly linked to negative emotions, positive emotions can moderate its effects. We also know that pictorial art and music improve mental health, and in particular that impressionist paintings can generate positive emotions. Finally, our App provides dual visual and auditory stimulation with the aim of triggering positive emotions, but this remains to be demonstrated. We therefore hypothesize that (1) observing and listening to musicalized Impressionist paintings can generate positive emotions, (2) the emotional effect is greater when the painting is associated with its music compared with simply observing the painting or listening to the music alone, and (3) the emotions triggered by observing and listening can change with age.

OBJECTIVES The primary objective is to characterize the emotional response during the presentation of Helen Mc Nicoll's painting Sunny September and Claude Monet's painting The Willows, by distinguishing 3 conditions: (1) contemplating each painting (visual stimulation), (2) listening to the original music composed from each painting (auditory stimulation), (3) contemplating and listening to the association of each painting with each specific music (bimodal stimulation), in young and elderly adults.

Secondary objectives were: - To determine whether the emotional profile is superimposable in terms of valence and arousal between visual and auditory stimulation of the original works (emotional congruence)

* To determine whether there is a synergistic effect in terms of valence and arousal when bimodal stimulation is used vs. two unimodal stimuli alone
* Determine which type of stimulation generates the strongest positive emotions in terms of valence and arousal
* Determine whether the order of stimuli (visual and auditory) has an effect on the elicitation of positive emotions and on their characteristics. - Evaluate whether emotional profiles vary according to the age group of participants
* Evaluate whether emotional profiles vary according to the gender of participants
* Evaluate whether the level of eco-anxiety prior to the aesthetic experience has an influence on emotional profiles following a nature-based aesthetic experience
* Evaluate whether the level of knowledge and engagement in the arts (visual as well as musical) has an influence on emotional profiles

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 35, or age 60 and over
* Sex and gender concordance
* No severe psychobehavioral or major neurocognitive disorders
* Have no severe visual or hearing impairment,
* Give written consent to participate in the study.

Exclusion Criteria:

* Participate in another concurrent experimental clinical study, to avoid interference with our study.
* Not understand written or spoken French or English.
* Identify as non-binary

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — In this protocol, we added an inclusion criterion on a match between the sex and gender of the participants. This limitation is important for controlling the key variable, which is the impact of gender and sex in the elicitation of emotions during stimulation.
  Gender differences in emotion characterization are documented through various measurement tools such as the Geneva Wheel of Emotions, the Self-Assessment Manikin (SAM) and electrodermal activity (EDA) which are used in our protocol. Studies using the SAM have shown that women tend to express more intense emotions, both positive and negative, than men, which is consistent with the greater emotional expressivity observed in women.
  Electrodermal activity, used to measure physiological arousal, also shows variations: men often show a higher electrodermal response, while women are more reactive in cooperative contexts.
  These results underline a gender-dependent modulation of emotions, influenced by biological and social factors.
Enrollment: 120 (Estimated)
Dates: Start 2025-01-22 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Physiological evaluation of emotions - electrodermal activity | Day 1
  Data acquisition of electrodermal activity (EDA) - tonic component (skin conductance level: SCL) and phasic component (skin conductance responses: SCR) EDA is the only index of sympathetic arousal induced by changes in emotional state, and is the only autonomic psychophysiological variable uncontaminated by parasympathetic activity.
Cognitive evaluation of emotions, discrete approach | Day 1
  Emotions using the discrete approach: thanks to the Geneva Emotions Wheel (GEW). Based on the circumplex theory of emotions, the GEW captures discrete and specific emotions in a way that is intuitive for participants and provides clear categories of emotions. This model was developed to represent and classify human emotions, drawing inspiration from the color wheel. It organizes emotions according to their intensity and relationship to each other, enabling clear visualization of interactions and oppositions between different emotions.
  After each stimulus (image, painting or music), the participant will be asked to indicate which main emotion he or she is feeling by selecting the appropriate segment of the wheel, and the level of intensity of the emotion felt by choosing the position on the corresponding circle.
Cognitive evaluation of emotions, dimensionnal approach | Day 1
  dimensional approach to emotions: using the Self Assessment Manikin (SAM). The SAM is a non-verbal tool that offers a continuous and graded assessment of emotions, which is useful for detecting fine nuances in emotional feelings. This scale measures three fundamental dimensions of emotion: valence (positivity/negativity), arousal, and control (dominance).
  After each stimulus, the participant will be asked to assess his or her feelings by choosing the figure that best represents his or her emotional experience on each of the three dimensions.
  Each dimension is represented by a series of five figures illustrating a linear progression. The user selects a figure that best represents his or her feelings on each dimension, or falls between 22 figures. This selection is then converted into a numerical score for each dimension. Typically, scores can range from 1 (extremely negative/not at all excited/low control) to 9 (extremely positive/very excited/high control).
Physiological evaluation of emotions - heart rate | Day 1
  pulse measurement by recording a photoplethysmogram and converting it to estimate heart rate.

SECONDARY OUTCOMES:
Level of engagement with music | up to 2 weeks before intervention day
  The MusEQ can be reliably used to explore the benefits of musical engagement in terms of cognitive and emotional regulation, engaged production, social connection and physical exercise. The scale comprises 32 questions to be answered on a 5-point Likert scale. These questions are divided into 6 subscales to assess 1/ daily behavior towards music, 2/ emotions, 3/ practice, 4/ consumption, 5/ behavior and 6/ preferences. Scores for each subscale are calculated by combining responses.
Level of commitment to art | up to 2 weeks before intervention day
  The VAIAK is a psychometric scale developed to assess two main aspects related to art: personal interest in art and level of artistic knowledge. Due to the complexity of the scale and the number of questions, we will only consider the part of the scale concerning the assessment of interest in art. This part of the scale measures a person's interest in and commitment to art. This includes aspects such as frequency of museum visits, interest in different art forms, and personal investment in artistic activities. This part is divided into 2 subscales: the first asking 8 questions to define the level of personal importance attached to art and the pleasure derived from these experiences on a 7-choice scale ranging from "not at all" to "enormously", the second asking 4 questions to define the frequency of interaction with art on a 7-choice scale ranging from "less than once a year" to "once a week or more".
Ecoanxiety level - Climate change | up to 2 weeks before intervention day
  Climate change anxiety scale (CCAS), developed by Clayton & Karaszia provides a 22-item measure of emotional reaction to climate change. It comprises four subscales, including cognitive and emotional impairment, functional impairment, personal experience of climate change and behavioral engagement. Each item is evaluated on a 5-point Likert scale ranging from "Never" to "Almost always" and worth 0 to 4 points, for a total score between 0 and 88. The higher the score, the greater the level of ecoanxiety. A low score indicates relatively low anxiety about climate change. The thresholds used in this project are: 0 to 22: low anxiety, 23 to 44: moderate anxiety, 45 to 66: high anxiety and 67 to 88: very high anxiety.
Ecoanxiety level - Environment issues | up to 2 weeks before intervention day
  Hogg ecoanxiety scale (HEAS-13): this 13-item scale measures anxiety in response to environmental problems and the climate crisis provides an ecological perspective on ecoanxiety. Each item is evaluated on a 4-point Likert scale ranging from "Never" to "Almost every day", and worth 0 to 3 points for a total score between 0 and 39. A low score indicates relatively low anxiety about environmental issues. The thresholds used in this project are: 0 to 12: low anxiety, 13 to 25: moderate anxiety and 26 to 39: high anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- CRIUGM, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided